CLINICAL TRIAL: NCT03590951
Title: Anesthetic and Obstetric Outcomes in Morbidly Obese Pregnant Patients Undergoing Cesarean Delivery: Retrospective Analysis of a Single Center Experience
Brief Title: Anesthetic and Obstetric Outcomes in Morbidly Obese Pregnancy and Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Other Study IDs: 1053583
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Morbid Obesity; Cesarean Section Complications; Pregnancy Related
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective chart review — A retrospective chart review was conducted to evaluate the effect of body mass index on obstetric, anesthetic and neonatal complications in patients who underwent cesarean section at our institution

SUMMARY:
Given that morbid obesity has been strongly associated with obstetric, neonatal and anesthetic complications, and that scarce reports have evaluated anesthetic and obstetric outcomes after cesarean delivery in morbidly obese patients; This study retrospectively analyzed anesthetic, obstetric and neonatal outcomes in morbidly obese pregnant patients who underwent cesarean delivery at Augusta University Medical Center, during a 2-year period (2015-2016).

DETAILED DESCRIPTION:
This study compared non-obese, obese and morbidly obese patients with respect to maternal, perinatal and anesthetic outcomes. Obstetric aspects included emergent procedure, estimated blood loss, obstetric complications, maternal disposition, length of stay and in-hospital mortality. Neonatal aspects included Apgar scores. Anesthetic aspects included anesthetic technique, intraoperative hemodynamic instability, failed regional anesthesia and anesthetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients who underwent cesarean section at Augusta University Medical Center.
* Patients older than 18 years.

Exclusion Criteria:

* Gestational age <37 weeks.
* Patients with chronic pain conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Term pregnant patients who underwent cesarean section between 2015 and 2016 at Augusta University Medical center.
Sampling Method: Non-Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Obstetric complications | From beginning to end of cesarean section (2 hours)
  Perioperative bleeding

SECONDARY OUTCOMES:
Anesthetic complications | From beginning to end of cesarean section (2 hours)
  Failed epidural
Neonatal complications | 1 and 5 minutes after delivery
  Apgar scores
Other anesthetic complications | From beginning to end of cesarean section (2 hours)
  Intraoperative hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros Perez, MD, Principal Investigator — Medical College of Georgia. Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No